CLINICAL TRIAL: NCT01811550
Title: Insights on Selected Procoagulation Markers and Outcomes in Stroke Trial (I-SPOT)
Brief Title: Study of Procoagulation Markers in Stroke Patients
Acronym: I-SPOT
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Neurological Emergencies Treatment Trials Network (NETT) (Network); University of Virginia (Other); University of Michigan (Other); Medical University of South Carolina (Other); Augusta University (Other)
Responsible Party: Sponsor
Other Study IDs: 11110979; 1U01NS079077-01A1 (NIH)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Hyperglycemia; Procoagulation Markers
MeSH Terms: conditions — Stroke; Hyperglycemia | interventions — Glycemic Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SHINE study subjects: Subjects enrolled in the SHINE trial who are not receiving intra-arterial therapy nor systemic anticoagulation; have no known moderate/severe hepatic insufficiency; have no known history of hypercoaguable or thrombotic condition; have INR =<1.5 (if known) at baseline and provide informed consent (self or LAR) will be enrolled in the I-SPOT study.
  Interventions: Other: Glycemic Control

INTERVENTIONS:
Other: Glycemic Control
  Other Names: Blood draw at 0 and 48 hours; Glycemic Control per SHINE protocol

SUMMARY:
The Insights on Selected Procoagulation Markers and Outcomes in Stroke Trial (I-SPOT): Response to Insulin Administration and Blood Glucose Control proposal is designed to accompany the Stroke Hyperglycemia Insulin Network Effort (SHINE) clinical trial, a Phase III multicenter, randomized, controlled trial planning to determine the efficacy and validate the safety of glycemic control in stroke patients. The SHINE trial will recruit 1,400 AIS patients with Type II diabetes mellitus (T2DM) and hyperglycemia, each receiving 3 days of hyperglycemia control with intravenous (IV) insulin therapy or control therapy with subcutaneous (SQ) insulin. The I-SPOT trial will recruit 315 SHINE patients. Blood coagulation marker levels will be measured before and at 48 hours after the start of treatment. Baseline and temporal changes in biomarkers levels will be compared between treatment groups.

Hypothesis: The decrease in levels of markers of blood coagulation will be greater in patients treated with IV insulin to reduce BG than in patients treated with SQ Insulin as the standard fashion.

Hypothesis: The decrease in levels of markers of blood coagulation will be greater in patients with than without favorable (SHINE) outcome (defined as the baseline stroke severity adjusted measure of functional ability at 90 days after AIS).

Hypothesis: Hyperglycemia control modulates the relationship between blood coagulation levels and functional outcome in T2DM patients after stroke. Patients treated with IV Insulin for hyperglycemia control with favorable (SHINE) outcome will have greater decreases in blood coagulation levels than either IV Insulin-treated patients without favorable outcome or SQ Insulin-treated with or without favorable outcomes at 90 days after AIS.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in SHINE study
* Ability to give Informed Consent (self or LAR)

Exclusion Criteria:

* Current or planned use of full dose anticoagulation from baseline to the 48 hour sample collection
* Known moderate or severe hepatic insufficiency (as defined by INR>1.5 if known or history of variceal bleeding or hepatic encephalopathy)
* Prior or concurrent thrombotic or hypercoagulable condition (Antiphospholipid antibody syndrome; Antithrombin III, Protein C or S deficiencies; Congenital or Inherited Factor deficiencies; sickle cell disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from participants in the SHINE trial.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2012-08; Primary Completion 2018-10 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
change in biomarker between patients with favorable versus unfavorable functional outcome | Randomization, 48 hours and 90 days

SECONDARY OUTCOMES:
Changes in biomarker levels between patients with versus without stroke recurrence at 90 days post stroke. | Randomization, 48 hours, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Nina T Gentile, M.D., Principal Investigator — Temple University
Locations (38):
- United States (38):
  - Banner University Medical Center, Tucson, Arizona
  - Long Beach Memorial Hospital, Long Beach, California
  - Ronald Regan Medical Center, Los Angeles, California
  - San Francisco General Hospital, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Detroit Receiving Hospital, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Kings County Hospital, Brooklyn, New York
  - SUNY Downstate University Hospital of Brooklyn, Brooklyn, New York
  - Kaleida Stroke Center, SUNY Buffalo, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Lincoln Medical and Mental Health Center, New York, New York
  - Summa Health System, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Wexner Medical Center, Columbus, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC - Mercy, Pittsburgh, Pennsylvania
  - UPMC - Presbyterian, Pittsburgh, Pennsylvania
  - UT Southwestern-Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern-Zale Lipshy University Hospital, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin